CLINICAL TRIAL: NCT01077089
Title: Effects of Transport on Patients With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rich Branson, M.D., Professor of Clinical-Geo, University of Cincinnati
Other Study IDs: Dorlac-2010-01
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; In-hospital transport
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transported TBI patients: Traumatically brain injured patients undergoing in-hospital transport.

SUMMARY:
Hospitalized patients are often moved from their rooms to other hospital locations, particularly imaging facilities. For patients with traumatic brain injury, such movements may raise the risk of secondary brain injuries. The purpose of this study is to monitor brain injured patients during transport and to measure the resulting changes in intracranial pressure. This will allow for documentation of the frequency of secondary injury and help in understanding their causes.

DETAILED DESCRIPTION:
Secondary insults, such as hypoxia and hypotension, may worsen a brain injury. We hypothesize that secondary brain insults may occur frequently during in-hospital transport in patients with traumatic brain injury (TBI). We additionally hypothesize that automated data collection devices used during transport could more reliably document the frequency of these events and help us to understand the causes. During transport of patients with TBI, intracranial pressure and arterial blood pressure will be continuously recorded to a monitor and saved for later analysis. Additional continuous measurements of pulse oximetry, end-tidal carbon dioxide, and mechanical ventilation settings will be made. The study will identify patients at risk for secondary insults, the etiology of these insults, and assist in development of a road map to prevent future incidents.

ELIGIBILITY:
Inclusion Criteria:

* presence of traumatic brain injury and intracranial pressure monitoring
* requiring mechanical ventilation
* presence of an indwelling arterial catheter for monitoring blood pressure
* Age of at least 18 years

Exclusion Criteria:

* Age less than 18 years
* diagnosis of brain death
* non-English speakers
* prisoners
* mentally ill persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events during transport. | Each transport event

SECONDARY OUTCOMES:
Incidence of elevated heart rate during transport. | Each transport event
Incidence of transport events during which SpO2 remains below 90% for 1 minute or longer | Each transport event
Transport events during which systolic blood pressure remains below 90 mmHg for 5 minutes or longer | Each transport event
Transport events during which mean arterial blood pressure remains below 60 mmHg for 5 minutes or longer | Each transport event
Transport events during which intracranial pressure exceeds 20 mmHg for 5 minutes or longer | Each transport event
Transport events during which cerebral perfusion pressure remains below 70 mmHg for 5 minutes or longer | Each transport event
Number of instances of physiological change that require caregiver intervention, such as ventilator manipulation or drug therapy | Each transport event

CONTACTS AND LOCATIONS:
Overall Officials: Warren A Dorlac, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Chesnut RM, Marshall LF, Klauber MR, Blunt BA, Baldwin N, Eisenberg HM, Jane JA, Marmarou A, Foulkes MA. The role of secondary brain injury in determining outcome from severe head injury. J Trauma. 1993 Feb;34(2):216-22. doi: 10.1097/00005373-199302000-00006. PMID 8459458
- [Background] Chesnut RM, Marshall SB, Piek J, Blunt BA, Klauber MR, Marshall LF. Early and late systemic hypotension as a frequent and fundamental source of cerebral ischemia following severe brain injury in the Traumatic Coma Data Bank. Acta Neurochir Suppl (Wien). 1993;59:121-5. doi: 10.1007/978-3-7091-9302-0_21. PMID 8310858
- [Background] Jeremitsky E, Omert L, Dunham CM, Protetch J, Rodriguez A. Harbingers of poor outcome the day after severe brain injury: hypothermia, hypoxia, and hypoperfusion. J Trauma. 2003 Feb;54(2):312-9. doi: 10.1097/01.TA.0000037876.37236.D6. PMID 12579057
- [Background] Manley G, Knudson MM, Morabito D, Damron S, Erickson V, Pitts L. Hypotension, hypoxia, and head injury: frequency, duration, and consequences. Arch Surg. 2001 Oct;136(10):1118-23. doi: 10.1001/archsurg.136.10.1118. PMID 11585502